CLINICAL TRIAL: NCT06487715
Title: Safety and Efficacy of Systemic Chemotherapy Plus PD-1 Inhibitor in Combination With Intraperitoneal Bevacizumab in Gastric Cancer With Peritoneal Metastasis
Brief Title: Safety and Efficacy of Systemic Chemotherapy Plus PD-1 Inhibitor in Combination With Bevacizumab in Gastric Cancer With Peritoneal Metastasis
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNION-GCPM
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer Peritoneal Metastases
MeSH Terms: interventions — Albumin-Bound Paclitaxel; S 1 (combination); sintilimab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Albumin-bound paclitaxel plus S1 and sintilimab in combination with Bevacizumab (Experimental): Intraperitoneal period: Albumin-bound paclitaxel plus S-1 combined with sintilimab (200 mg, d1) and bevacizumab (7.5 mg/m2, d1) intraperitoneally, 3-week cycle, 2 cycles; Maintenance period: Albumin-bound paclitaxel plus S-1 combined with sintilimab (200 mg, d1) and bevacizumab (7.5 mg/m2, d1) intravenously, 3-week cycle
  Interventions: Drug: albumin-bound paclitaxel (260 mg/m2, d1); Drug: S-1; Drug: sintilimab; Drug: bevacizumab

INTERVENTIONS:
Drug: albumin-bound paclitaxel (260 mg/m2, d1) — 260 mg/m2, d1)
Drug: S-1 — 80 mg/m2, d1-14
Drug: sintilimab — 200 mg, d1
Drug: bevacizumab — First two cycles : intraperitoneally 7.5 mg/m2 Maintenance period: intravenously 7.5 mg/m2

SUMMARY:
It is an open label, phase II study involved receiving albumin-bound paclitaxel plus S-1 combined with sintilimab and bevacizumab in patients with gastric cancer peritoneal metastasis.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years patients histologically or cytologically confirmed the presence of GC or gastroesophageal junction tumor with PM (HER2 negative). The ECOG performance status is 0-1 and the expected survival time is more than 3 months. Did not receive any therapy for GC within the last six months (chemotherapy, radiation therapy, or both).

Exclusion Criteria:

* Principal exclusion criteria: The obstruction of the cardia and pylorus affects the patient's eating and gastric emptying, or has difficulty swallowing tablets. HER2-positive GC and gastroesophageal junction tumors. Subject with other malignancies, except for non-melanoma skin cancer or in-situ cervical carcinoma under adequate treatment, or other treated malignancies without evidence of recurrence for 5 years. Previously received the following therapies: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs that stimulate or co-inhibit T cell receptors (eg, CTLA-4, OX-40, CD137). Received systemic treatment with Chinese medicines or immunomodulatory drugs (including thymosin, interferon, interleukin, except for local use to control pleural effusion) with anti-tumor indications within 2 weeks before the first administration; Active autoimmune disease requiring systemic therapy (eg, disease-modifying drugs, glucocorticoids, or immunosuppressants) occurred within 2 years prior to first dose; Replacement therapy (such as thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency, etc.) is not considered systemic therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | 1 year

SECONDARY OUTCOMES:
Progression free survival | 1 year
Ascites drainage-free survival | 1 year
Objective Response Rate | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No